CLINICAL TRIAL: NCT07388680
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase II/III Clinical Trial on the Efficacy and Safety of Hydronidone Capsules in the Treatment of Radiation-induced Lung Injury With or Without Immune-related Pneumonia
Brief Title: Hydronidone Capsules in the Treatment of Radiation-induced Lung Injury With or Without Immune Pneumonia
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beijing Continent Pharmaceutical Co, Ltd. (Industry)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KDN-F647-202401
Record Dates: First submitted 2025-11-17; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Radiation-induced Lung Injury; Immune-related Pneumonia
Keywords: Radiation-induced lung injury; Immune-related pneumonia; RILI; CIP
MeSH Terms: interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-dose group (Experimental): Pirfenidone Capsules (Low-dose group: 400 mg, TID)
  Interventions: Drug: Pirfenidone Capsules （400 mg）
- High-dose group (Experimental): Pirfenidone Capsules (High-dose group: 600 mg, TID)
  Interventions: Drug: Pirfenidone Capsules（600mg）
- Placebo group (Placebo Comparator): Pirfenidone Capsules（0mg，TID）
  Interventions: Drug: Pirfenidone Capsules（0mg）

INTERVENTIONS:
Drug: Pirfenidone Capsules （400 mg） — Low-dose group:400 mg, TID
  Arms: Low-dose group
Drug: Pirfenidone Capsules（600mg） — Pirfenidone Capsules（600mg，TID）
  Arms: High-dose group
Drug: Pirfenidone Capsules（0mg） — Placebo（0mg，TID）
  Arms: Placebo group

SUMMARY:
Radiation-induced lung injury (RILI) is one of the most common thoracic-radiotherapy complications, with an incidence as high as 31.4 %. Multiple studies have shown that RILI can adversely affect patient prognosis by disrupting treatment schedules. Moreover, the widespread clinical use of immune-checkpoint inhibitors (ICIs) has further increased pulmonary toxicity when radiotherapy (RT) is combined with ICIs. Checkpoint-inhibitor-related pneumonitis (CIP)-i.e., immune-mediated lung injury-may necessitate permanent discontinuation of ICIs, diminish survival benefit, and, in severe cases, directly threaten life. The diagnosis of both RILI and CIP is based on an integrated assessment of subjective symptoms and imaging findings.RILI typically occurs 1-3 months after completion of radiotherapy, whereas CIP may emerge at any point during treatment. The two entities share similar clinical presentations: fever, dry cough, chest tightness, dyspnoea, and pleuritic chest pain. Computed tomography (CT) is the most sensitive imaging modality. Pulmonary-function testing is another routinely used clinical metric; vital capacity, total lung capacity, forced expiratory volume in 1 s (FEV₁), and diffusing capacity of the lung for carbon monoxide (DLCO) may all decline, with DLCO being the most sensitive parameter. In advanced cases, arterial oxygen and carbon-dioxide tensions may also deteriorate.Currently, RILI is managed empirically with systemic corticosteroids and supportive care; however, this approach yields limited improvement in diffusing capacity or ventilatory function, and its ability to prevent radiation-induced pulmonary fibrosis (RPF) remains undefined. Corticosteroids also remain the mainstay of CIP therapy. Pirfenidone, a potent cytokine inhibitor, attenuates fibroblast activity by reducing production of transforming growth factor-β1 (TGF-β1), platelet-derived growth factor (PDGF), and fibroblast growth factor (FGF), thereby suppressing fibroblast proliferation and extracellular-matrix collagen synthesis. Pre-clinical efficacy studies have demonstrated robust anti-inflammatory, anti-oxidant, and anti-fibrotic effects in the lung.Because RILI and pneumonitis arising from combined radio-immunotherapy are often indistinguishable in clinical practice, and because both share pathogenetic features with idiopathic pulmonary fibrosis (IPF), the investigators initiated this phase II/III trial to address the unmet medical need for effective therapy. Building on prior pre-clinical and clinical data, the study aims to establish the optimal dose of pirfenidone capsules for RILI with or without concomitant CIP and to confirm efficacy and safety.Phase II (dose-finding): The study consists of a screening period (Day -28 to Day -1), a 168-day treatment-observation period (Day 1-Day 168), a safety follow-up (28 ± 7 days after the last dose), and subsequent disease-progression and survival follow-up. Ninety subjects with RILI, with or without CIP, who meet all eligibility criteria will be randomly assigned 1:1:1 to low-dose pirfenidone (400 mg TID), high-dose pirfenidone (600 mg TID), or matching placebo.Phase III (confirmatory): The dose of pirfenidone capsules for phase III will be determined jointly by the sponsor and investigators based on accumulated efficacy and safety data. The trial structure mirrors phase II: screening (Day -28 to Day -1), 168-day treatment-observation (Day 1-Day 168), safety follow-up (28 ± 7 days after the last dose), and disease-progression and survival follow-up. Eligible subjects with RILI ± CIP will be randomized 1:1 to receive either pirfenidone capsules (400 mg or 600 mg TID, taken with meals) or identical placebo. After completion of the 28-day post-treatment follow-up, all phase III participants will enter an extension phase for long-term survival assessment every 3 months (± 7 days).

ELIGIBILITY:
Inclusion Criteria:

* The subjects must meet all the following inclusion criteria to be enrolled in this study:
* Voluntary signing of the informed consent form, and being capable of understanding and signing the informed consent form before the study.
* Age 18 to 75 years (inclusive of 18 and 75), with no gender restrictions.
* Malignant tumors diagnosed by pathological histology/cytology, and having received radiotherapy to the chest.
* According to the Common Terminology Criteria for Adverse Events (CTCAE) v5.0 standard, diagnosed by the investigator as clinical RILI grade 2-3 with or without CIP. For those with CIP, the investigator determines that only hormone treatment is required.
* At the time of enrollment, 40% ≤ DLCO as a percentage of the predicted value < 80% (mild to moderate lung diffusion function impairment).
* The course of radiation-induced lung injury is less than 2 months.
* If receiving radiation-induced lung injury-related treatment (including glucocorticoids, antibiotics, etc.) at the time of enrollment, the types and doses of medication must remain stable within 2 weeks before enrollment, and the hormone medication does not exceed 4 weeks.
* At the time of enrollment, the investigator assesses that the subjects can take oral administration of the investigational drug.
* Eastern Cooperative Oncology Group score (ECOG) 0-2.
* Expected survival period ≥ 6 months.
* The functional level of major organs meets the following standards:

  1. Blood routine examination: Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count (PLT) ≥ 75 × 109/L or hemoglobin (Hb) ≥ 90 g/L;
  2. Biochemical examination: Total bilirubin (TBIL), blood urea nitrogen (BUN), and creatinine (Cr) ≤ 1.5 upper limit of normal value (ULN), or creatinine clearance rate ≥ 50 mL/min; alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 2.0 ULN.

     * Creatinine clearance rate = [(140 - age) × weight (kg)] / [0.818 × Scr (umol/L)] (for females × 0.85)
* For all fertile women, the serum pregnancy test within 7 days before the first administration must be negative, and fertile male and female subjects must agree to use reliable contraceptive methods (hormonal or barrier method or abstinence) with their partners during the entire study period and at least 6 months after the last use of the investigational drug.

Exclusion Criteria:

* Subjects with Child-Pugh grade C at the time of enrollment or with severe liver diseases such as liver failure, hepatic encephalopathy, etc.
* Subjects who have had Stevens-Johnson syndrome, toxic epidermal necrolysis (TEN), drug eruption with eosinophilia and systemic symptoms (DRESS), or severe skin diseases in the past or currently;
* Subjects who have other diseases that the investigator deems unsuitable for participation in this study during the screening process.
* Subjects with active untreated brain metastases or meningeal metastases; for subjects with treated central nervous system (CNS) metastases, if the symptoms are controlled for at least 4 weeks, they are eligible for enrollment;
* Subjects who have a second malignancy that requires concurrent systemic cytotoxic chemotherapy, investigational treatment or biological therapy (such as anti-cytotoxic T lymphocyte-associated protein 4 [CTLA4] or human epidermal growth factor receptor 2 [HER2] monoclonal antibodies), but are allowed to enroll if they have a second malignancy that only requires hormone therapy (such as gonadotropin-releasing hormone [LHRH] agonists, tamoxifen, etc.);
* Subjects with a history of human immunodeficiency virus (HIV) infection, or positive HIV antibodies or suspected HIV infection.
* Subjects who cannot discontinue tetracycline antibiotics (such as doxycycline, minocycline, etc.) within 14 days before screening or during the study.
* Subjects who the investigator deems unable to follow the testing procedures (such as being unable to tolerate the interruption of assisted oxygen supply during pulmonary function tests).
* Subjects who have used or are to use drugs that may have preventive and/or therapeutic effects on radiation pneumonitis within 1 month before screening or during the study, such as pentoxifylline, angiotensin-converting enzyme inhibitors, berberine, ursolic acid, statins, nicorandil, stem cells, interferon-γ, penicillamine, etc.;
* Subjects who have used nintedanib or high-dose acetylcysteine within 1 month before randomization;
* Subjects who have used known or judged by the investigator to be beneficial to lung injury Chinese herbal medicines or other substances during the 1 month before randomization;
* Subjects who have received or been exposed to live vaccines or attenuated live vaccines or plan to receive live vaccines or attenuated live vaccines (except anti-tumor treatment live vaccines) during the study;
* Subjects who have used drugs that are strong inhibitors or inducers of cytochrome CYP1A2, CYP2C9, CYP2C19, CYP2D6, CYP2E1 within 1 month before screening or during the study;
* Female subjects who are breastfeeding at the time of screening or male subjects whose partner is planning to get pregnant during the study.
* Subjects with known mental disorders that may affect the study assessment or with poor compliance.
* Subjects who are allergic to any active ingredients of this drug or its excipients (such as lactose) or lactose intolerant.
* Subjects who had severe trauma or received surgery within 1 month before screening or during the study, or who plan to undergo surgery during the study.
* Subjects who, according to the investigator's judgment, have other serious systemic diseases or laboratory test abnormalities or other reasons that make them unsuitable for participating in this clinical trial.
* Subjects who plan to participate in other drug clinical trials during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Phase II and Phase III: The absolute value of the change in the predicted percentage of lung carbon monoxide diffusion capacity (DLCO% predicted) from the baseline at week 24. | At the 24th week of the experiment
  DLCO% is a core indicator for evaluating pulmonary gas exchange function, reflecting the efficiency of oxygen transfer from the alveoli into the bloodstream. It is crucial for the diagnosis and prognosis of interstitial lung disease, pulmonary vascular disease, and similar conditions. DLCO% = measured diffusing capacity of the lung for carbon monoxide ÷ predicted value × 100%. Absolute value change refers to the direct difference between two consecutive measurements (for example, a decrease from 65% to 55% represents an absolute value change of -10%).

SECONDARY OUTCOMES:
Phase II and Phase III: The absolute values of the changes in DLCO% at weeks 2, 4, 8, and 16 compared to the baseline. | At weeks 2, 4, 8 and 16 of the trial
Phase II and III: Compared with the baseline, the changes in the measured values of pulmonary carbon monoxide diffusion capacity (DLCO) (in units of liters [L]) at weeks 2, 4, 8, 16, and 24. | At weeks 2, 4, 8,16 and 24 of the trial
Phase II and Phase III: Changes in forced vital capacity (FVC) (in liters) from baseline at weeks 2, 4, 8, 16, and 24. | At weeks 2, 4, 8,16 and 24 of the trial
Phase II and Phase III: The absolute value changes of forced vital capacity as a percentage of the predicted value (FVC%) from baseline at weeks 2, 4, 8, 16, and 24. | At weeks 2, 4, 8,16 and 24 of the trial
Phase II and Phase III: Changes in forced expiratory volume in one second (FEV1) (in liters) from baseline at weeks 2, 4, 8, 16, and 24. | At weeks 2, 4, 8,16 and 24 of the trial
Phase II and Phase III: The absolute value of the change in forced expiratory volume in one second as a percentage of the predicted value (FEV1%) from baseline at weeks 2, 4, 8, 16, and 24. | At weeks 2, 4, 8,16 and 24 of the trial
Phase II and Phase III: Changes in FEV1/FVC from baseline at weeks 2, 4, 8, 16, and 24. | At weeks 2, 4, 8,16 and 24 of the trial
Phase II and Phase III: Changes in the St. George's Respiratory Questionnaire (SGRQ) scores from baseline at weeks 4, 8, 16, and 24. | At weeks 4, 8,16 and 24 of the trial
  The St. George's Respiratory Questionnaire (SGRQ) score is the standard instrument for assessing health-related quality of life in patients with chronic airway diseases. It comprises 76 items grouped into three domains-symptoms, activity, and disease impact. Each domain score and the overall total score are scaled from 0 to 100: 0 denotes "complete absence of symptoms or limitation," whereas 100 indicates "maximal severity." Higher scores signify a greater adverse effect of the disease on daily life.
Phase II and Phase III: Changes in cough score from baseline at weeks 2, 4, 8, 16, and 24. | At weeks 2, 4, 8,16 and 24 of the trial
  The cough score is a subjective instrument that quantifies the frequency, intensity, and disruptive impact of cough on daily activities and sleep into a 0-10-point or 0-100-mm scale; zero denotes complete absence of cough, and higher values indicate increasing symptom severity.
Phase II and Phase III: Changes in the Modified Medical Research Council Dyspnea Scale (mMRC) score at weeks 2, 4, 8, 16, and 24 compared to the baseline. | At weeks 2, 4, 8,16 and 24 of the trial
  The Modified Medical Research Council Dyspnea Scale (mMRC) is a five-level instrument that rapidly quantifies the extent to which breathlessness limits physical activity; higher grades indicate greater disability.
Phase II and Phase III: Compared with the baseline, the changes in computed tomography (CT) imaging scores at weeks 4, 8, 16, and 24 | At weeks 4, 8,16 and 24 of the trial
  CT imaging score is a standardized method that converts anatomical or functional features observed on CT scans into quantifiable numerical values, used for disease diagnosis, staging, treatment response monitoring, or prognostic assessment.Referring to the HRCT scoring system, the scores were assigned by imaging experts after consensus , with higher values generally indicating more severe disease.
Phase II and Phase III: The proportion of subjects with CIP at baseline who discontinued immunotherapy and experienced immune reactivation during the study period. | Within 24 weeks
Phase II and Phase III: The proportion of subjects whose lung injury grade decreased by at least one level compared to the baseline at week 24. | Within 24 weeks
  According to the Common Terminology Criteria for Adverse Events, Version 5.0, pulmonary injury is graded, with higher grades indicating more severe symptoms.
Phase II and Phase III: The proportion of subjects achieving a lung injury level of ≤ 1 at the 24th week compared to the baseline. | Within 24 weeks
  According to the Common Terminology Criteria for Adverse Events, Version 5.0, pulmonary injury is graded, with higher grades indicating more severe symptoms.
Phase II and Phase III: The time required for the subjects to first achieve a lung injury level of ≤ 1. | Within 24 weeks
  According to the Common Terminology Criteria for Adverse Events, Version 5.0, pulmonary injury is graded, with higher grades indicating more severe symptoms.
Phase II and Phase III: The proportion of subjects who experienced their first acute pulmonary deterioration or died for any reason within 24 weeks of treatment. | Within 24 weeks
  Acute pulmonary deterioration is defined as the unexplained worsening or new onset of cough, dyspnea, hypoxia, or pneumonia from the completion of initial treatment up to Week 24, persisting for >4 days, with chest CT showing new or increased diffuse pulmonary infiltrates in the absence of pneumothorax or pleural effusion, and after exclusion of pneumonia, congestive heart failure, pulmonary embolism, or cancer progression. Pulmonary deterioration occurring within the first 2 weeks after initial treatment is not counted toward the endpoint, allowing full resolution of initial symptoms.
Phase II and Phase III: Analyze the blood drug concentration of pirfenidone capsules, evaluate the steady-state blood drug trough concentration for individual patients and each group of people at specific treatment time poin | on days 1, 14, 28, 56, 112, and 168 of the trial
Phase II and Phase III: Analyze the blood drug concentration of pirfenidone capsules, evaluate the PopPK characteristics for individual patients and each group of people at specific treatment time poin | on days 1, 14, 28, 56, 112, and 168 of the trial
Phase II and Phase III: Adverse events/serious adverse events (AE/SAE). | Within 24 weeks
  Adverse Event (AE) refers to any untoward and unintended medical occurrence experienced by a trial participant during treatment or clinical investigation, regardless of causal relationship to the investigational product. Serious Adverse Event (SAE) is a subset of AE that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, causes persistent or significant disability/incapacity, leads to congenital anomaly/birth defect, or is judged medically important by the investigator.
  According to the Common Terminology Criteria for Adverse Events, Version 5.0, pulmonary injury is graded, with higher grades indicating more severe symptoms.
Phase II and Phase III:Number of participants with abnormal ECG readings | At weeks 2, 4, 8,16 and 24 of the trial
Phase II and Phase III: vital signs( blood pressure). | At weeks 2, 4, 8,16 and 24 of the trial
  Record patient's systolic and diastolic blood pressure
Phase II and Phase III: vital signs(pulse rate). | At weeks 2, 4, 8,16 and 24 of the trial
Phase II and Phase III: vital signs(body temperature). | At weeks 2, 4, 8, 16 and 24 of the trial
Phase II and Phase III: vital signs( respiratory rate data). | At weeks 2, 4, 8, 16 and 24 of the trial
Phase II and Phase III: laboratory tests（complete blood count). | At weeks 2, 4, 8, 16 and 24 of the trial
Phase II and Phase III: Number of participants with abnormal urinalysis | At weeks 2, 4, 8, 16 and 24 of the trial
Phase II and Phase III: Number of participants with abnormal laboratory tests results (blood biochemistry) | At weeks 2, 4, 8, 16 and 24 of the trial
Phase II and Phase III: Number of participants with abnormal laboratory tests results (coagulation function) | At weeks 2, 4, 8, 16 and 24 of the trial
Phase II and Phase III: laboratory tests( pregnancy test for safety assessment). | At weeks 2, 4, 8, 16 and 24 of the trial

OTHER OUTCOMES:
Phase II and Phase III : Analysis of the correlation between cytokines and efficacy and safety. | on days 1, 28, and 168 of the trial
  Flow cytometry was employed to analyze the correlation between pirfenidone and immune-cell subsets (CD8⁺ T cells, CD4⁺ T cells, regulatory T cells [Treg], and macrophages).

CONTACTS AND LOCATIONS:
Overall Officials: Ming Chen, Principal Investigator — Sun Yat-sen University
Locations (36):
- China (36):
  - Anhui Provincial Chest Hospital, Hefei, Anhui
  - Chinese Academy of Medical Sciences Cancer Hospital, Beijing, Beijing Municipality
  - Affiliated Hospital of Fujian Medical University, Xiehe Branch, Fuzhou, Fujian
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Lanzhou University First Hospital, Lanzhou, Gansu
  - Foshan First Hospital, Foshan, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Panyu Central Hospital Affiliated to Guangzhou Medical University, Guangzhou, Guangdong
  - Southern Medical University - Southern Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Gaozhou People's Hospital, Maoming, Guangdong
  - Chinese Academy of Medical Sciences Cancer Hospital Shenzhen Branch, Shenzhen, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Affiliated Hospital of Guangdong Medical UniversityAffiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Zhongshan People's Hospital, Zhongshan, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - The Second Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Hebei University Affiliated Hospital, Baoding, Hebei
  - Anyang City Cancer Hospital, Anyang, Henan
  - Henan Provincial Cancer Hospital, Zhengzhou, Henan
  - Hubei Provincial Cancer Hospital, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xuzhou Medical University Affiliated Hospital, Xuzhou, Jiangsu
  - Gansu Provincial Cancer Hospital, Gansu, Lanzhou
  - Jining First People's Hospital, Jining, Shandong
  - Fudan University Cancer Hospital, Shanghai, Shanghai Municipality
  - Shanghai Chest HospitalShanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Sichuan Provincial Cancer Hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Hunan Provincial Cancer HospitalHunan Provincial Cancer Hospital, Changsha, Wuhan
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial Cancer HospitalZhejiang Provincial Cancer Hospital, Hangzhou, Zhejiang
  - Taizhou Cancer Hospital, Taizhong, Zhejiang